CLINICAL TRIAL: NCT06646926
Title: The Immediate and 24-hour Effects of Body Tempering Versus Foam Rolling on Lower Extremity Muscular Power During the Vertical Jump and Standing Long Jump Tests
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Matthew Geary, Clinical Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00139385
Record Dates: First submitted 2024-10-04; First posted 2024-10-17 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Lower Extremity Muscular Power Performance Output
Keywords: lower extremity; muscle power; body tempering; foam rolling; myofascial release

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Body Tempering (Experimental): Participant will be positioned prone on the Body Tempering Ab Mat with their feet hanging off the end of the mat. The body tempering intervention will be applied by the same investigator for all trials. The body tempering device will be applied dynamically to each participant for 4 minutes, with the device placed on both participants' lower extremities at the same time. First, the examiner will set a timer for two minutes and begin rolling one 80-pound body tempering device along the participant's gastrocnemius-soleus complex at a rate of 30 beats per minute, traveling from the Achilles tendon (medial malleolus) to the inferior aspect of the popliteal fossa, indicated by fibular head. The participant will then take thirty seconds to transition to a supine position and receive tempering with an 80-pound tempering device along their middle to distal quadriceps, set a timer for 2 minutes.
  Interventions: Other: Body tempering
- Foam rolling self-myofascial release (Active Comparator): Participants will be instructed via standardized script to perform self-myofascial release (SMR) on their gastrocnemius-soleus complex and quadriceps muscles. The first SMR sequence will be performed by having the participant place the foam roller behind both calves, beginning the roll at the medial malleolus and ending at the inferior aspect of the popliteal fossa, indicated by the fibular head. The participant will perform this for two minutes, rolling at a tempo of 30 beats per minute. Next, the participant will take thirty seconds to transition to a prone position, placing the foam roller just distal to the hip crease, just inferior to the AIIS, and rolling inferiorly to the area just proximal to the most superior aspect of the patella. This self-release sequence will be performed for two minutes at a tempo of 30 beats per minute. The total time should be four minutes, matching the total time of the experimental intervention group.
  Interventions: Other: Foam rolling self-myofascial release

INTERVENTIONS:
Other: Body tempering — Participant will be positioned prone on the Body Tempering Ab Mat with their feet hanging off the end of the mat. The body tempering intervention will be applied by the same investigator for all trials. The body tempering device will be applied dynamically to each participant for 4 minutes, with the device placed on both participants' lower extremities at the same time. First, the examiner will set a timer for two minutes and begin rolling one 80-pound body tempering device along the participant's gastrocnemius-soleus complex at a rate of 30 beats per minute, traveling from the Achilles tendon (medial malleolus) to the inferior aspect of the popliteal fossa, indicated by fibular head. The participant will then take thirty seconds to transition to a supine position and receive tempering with an 80-pound tempering device along their middle to distal quadriceps, set a timer for 2 minutes.
  Arms: Body Tempering
Other: Foam rolling self-myofascial release — Participants will be instructed via standardized script to perform self-myofascial release (SMR) on their gastrocnemius-soleus complex and quadriceps muscles. The first SMR sequence will be performed by having the participant place the foam roller behind both calves, beginning the roll at the medial malleolus and ending at the inferior aspect of the popliteal fossa, indicated by the fibular head. The participant will perform this for two minutes, rolling at a tempo of 30 beats per minute. Next, the participant will take thirty seconds to transition to a prone position, placing the foam roller just distal to the hip crease, just inferior to the AIIS, and rolling inferiorly to the area just proximal to the most superior aspect of the patella. This self-release sequence will be performed for two minutes at a tempo of 30 beats per minute. The total time should be four minutes, matching the total time of the experimental intervention group.
  Arms: Foam rolling self-myofascial release

SUMMARY:
The goal of this clinical trial is to examine the effects of body tempering on healthy volunteers between the ages of 18-39. The main question it aims to answer is will the intervention have an impact on immediate or 24-hour measures of lower extremity power as measured by the:

vertical jump test? standing long jump test? Researchers will compare an alternate intervention of foam rolling self-myofascial release to see if any changes in jump test performance are comparable.

Participants will perform a brief warm-up followed by baseline performance of the two jump tests (5 repetitions each). Participants will be randomized into one of two groups: either application of the body tempering intervention or performance of self-myofascial release via foam rolling. Following the intervention, participants will be asked to perform 3 repetitions of each outcome measure (jump test); participants will be asked to return 24 hours later where they will guided through the same warm-up as the day prior and will again perform 5 repetitions of each jump test.

DETAILED DESCRIPTION:
All procedures will take place on the first floor of the Solomon Blatt Physical Education Center in Lab Rooms 104, 105, 108, the first-floor hallway, and the first floor stairwell. Data collection will be performed in the fall 2024 and spring 2025, data analysis will be performed in the fall of the same year, and research defense will be performed in the fall of the same year. Participants will be assigned to either a body tempering or self-myofascial release (SMR) group via simple randomization for sex, with at least fifteen participants being placed into each group. Informed consent and IRB approval will be obtained prior to data collection. The group assignment of each participant will be known to the lead investigators who will be a licensed physical therapist and two examiners, one coordinating the warmup and the other performing the intervention. The data collector will remain blind to group assignments. Each participant will be required to sign an informed consent form and will be allowed to opt out of future data collection or to no longer participate in the study at any time, without any negative consequences to the participant, as they will not be receiving any compensation for participation.

Participants, ages 18-39, will be recruited via word-of-mouth, flier, and email on the University of South Carolina campus. Prior to the intervention's application, each subject will sign an informed consent form after a proper explanation by the primary investigator of the study's intent and the possibility of injury. To ensure the safety of the participants, each participant will be required to fill out a participant information form to screen for possible contraindications which include the following: history of knee or hip injury, hypertension, thrombophlebitis, inflammation, myositis ossificans, osteomyelitis, open wounds, unhealed fractures, hematoma, hemophilia, pregnancy, cancer, burns or skin grafts, varicose veins, synovitis, currently taking any anticoagulation medications, rheumatoid arthritis, osteoporosis or any other condition that would prevent subject participation. Once completed, the primary investigator will review each subject form and make the final decision as to include or exclude the individual(s) from the study. Lastly, to preserve subject privacy, each subject will be assigned a participant number to be used for reference during data entry and analysis.

Included in all announcements, fliers and emails, participants will be informed that they need to wear athletic attire to be included in the study. If the participants are unable to wear the required attire, they will be provided with a pair of paper shorts which can be disposed of after their participation in the 24-hour retest has concluded.

After it has been determined that the participant meets the eligibility criteria, the participant will be instructed to perform a standardized warm-up to limit variability among their physical readiness to participate. The warm-up will include a three-minute jog at 50% of their perceived maximum exertion, five seconds of high knees (hip flexion to ~90 degrees) at 50% of their perceived maximum exertion, and five seconds of butt-kicks (maximal knee flexion) at 50% of their perceived maximum exertion. After completing the warm-up, the participant will be instructed to rest for two minutes to decrease any accumulated fatigue. After the allotted two minutes of rest, participants will then move to take baseline measurements on the vertical jump and broad jump respectively with an investigator (AC) present to perform measurements. After performing baseline measurements, participants will return to Blatt PE Center Room 104 to be randomly allocated into intervention group by the investigator performing intake.

For the intervention group, the participant will be positioned in the prone position on the Body Tempering Ab Mat, purchased from https://roguefitness.com, with their feet hanging off the end of the mat. The body tempering intervention will be applied by the same investigator for all trials. The body tempering device will be applied dynamically to each participant for four minutes, with the device placed on both participants' lower extremities at the same time. First, the examiner will set a timer for two minutes and begin rolling one 80-pound body tempering device along the participant's gastrocnemius-soleus complex at a rate of 30 beats per minute, as indicated by the Pro Metronome iPhone© Version 4.2 application, traveling from the Achilles tendon (medial malleolus) to the inferior aspect of the popliteal fossa, indicated by fibular head. The participant will then take thirty seconds to transition to a supine position as indicated for dynamic tempering along bilateral quadriceps in the Body Tempering™ Course Manual. The examiner will place the 80-pound body tempering device along participants' middle to distal quadriceps, set a timer for 2 minutes, and dynamically temper from one hand width (as measured by the participants hand width) distal to the hip crease to just proximal to the most superior aspect of the patella at a rate of 30 beats per minute.

The control participants will be instructed via standardized script to perform self-myofascial release (SMR) on their gastrocnemius-soleus complex and quadriceps muscles. The first SMR sequence will be performed by having the participant place the foam roller behind both calves, beginning the roll at the medial malleolus and ending at the inferior aspect of the popliteal fossa, indicated by the fibular head. The participant will perform this movement for two minutes, rolling at a tempo of 30 beats per minute, being provided the Pro Metronome iPhone© Version 4.2 application. Next, the participant will take thirty seconds to transition to a prone position, placing the foam roller just distal to the hip crease, just inferior to the AIIS, and rolling inferiorly to the area just proximal to the most superior aspect of the patella. This self-release sequence will be performed for two minutes at a tempo of 30 beats per minute. The total time should be four minutes, matching the total time of the intervention group.

The vertical jump assessment will be performed according to the protocol used by Sayers and colleagues. Participants will cover the fingers of their dominant hand with chalk and stand beside a wall, descend into a squat with a 90-degree knee bend, and, after pausing for two seconds, will jump as high as they are able, reaching up with their dominant hand and placing a mark on the wall. Participants will perform this sequence five times. However, only the last three trials being recorded, which will be unknown to participants. The greatest value obtained from the trials will be used to calculate lower extremity power using the regression formula produced by Sayers and colleagues (Peak Power (W) = (60.7) × (jump height [cm]) + 45.3 × (body mass [kg]) - 2055). Rest intervals will be the amount of time it takes to complete the measurement for each trial.

Similarly, the standing long jump assessment (SLJ) assessment will be performed for five trials with the best performance on the three experimental trials used to determine lower extremity power. The SLJ will be performed like the protocol used by Mann and colleagues with participants performing horizontal jumps as far as they can and measuring the distance from the start point to the back of the subject's backmost heel. The subject must maintain their balance after landing for the trial to be counted. The farthest distance jumped will then be used to calculate power through the regression formula created by Mann and colleagues (Power [W] = 32.49·SLJ [cm] + 39.69·Wt [kg] - 7,608). Rest time between trials will be the amount of time it takes to measure the distance the subject jumped.

When the participants return for the 24-hour reassessment, they will be guided through the standardized warmup and retested with the vertical jump assessment and the standing long jump. Following the last measure of both sessions, participants will complete a Global Rating of Change scale consisting of a one-question prompt and eleven answer choices to gauge their perception of change in performance after receiving the intervention. The prompts are placed on a scale from -5 (Performed worse) to +5 (Performed better) and 0 (Stayed the same). The Global Rate of Change Scale will be given at the end of sessions 1 and 2 and will be completed the same to determine how much the subject's perceived effectiveness of body tempering and foam rolling. Each intervention group will receive a Global Rating of Change Scale specific to the intervention they received to ensure there is no confusion with the prompt.

To measure the difference between interventions (Body tempering and Foam Rolling) and different time points (Pre-, Post-, and 24-post intervention) repeated measures ANOVAs will be performed separately for the vertical jump and standing long jump assessments. Post hoc analysis will be used to determine the variables that caused any change seen in the experiment. Additionally, effect sizes will be calculated to determine the overall significance of any differences seen between experimental groups using Cohen's d. The effect size will be defined as large (d>0.8), medium (d=0.5), or small (d=0.2). A Mann-Whitney U test will also be run to determine the difference in Global Rate of Change scores between interventions and time points in our experiment.

ELIGIBILITY:
Inclusion Criteria:

• Healthy subjects age 18-39 years old

Exclusion Criteria:

* History of knee or hip injury,
* Hypertension
* Thrombophlebitis
* Inflammation
* Myositis ossificans
* Osteomyelitis
* Open wounds
* Unhealed fractures
* Hematoma
* Pregnancy
* Cancer
* Burns or Skin grafts
* Varicose veins
* Synovitis
* Currently taking any anticoagulation medications
* Rheumatoid arthritis
* Osteoporosis

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
vertical jump test | From enrollment to the end of follow up assessment at 24 hours
  The vertical jump assessment will be performed according to the protocol used by Sayers and colleagues. Participants will cover the fingers of their dominant hand with chalk and stand beside a wall, descend into a squat with a 90-degree knee bend, and, after pausing for two seconds, will jump as high as they are able, reaching up with their dominant hand and placing a mark on the wall. Participants will perform this sequence five times. However, only the last three trials being recorded, which will be unknown to participants. The greatest value obtained from the trials will be used to calculate lower extremity power using the regression formula produced by Sayers and colleagues (Peak Power (W) = (60.7) × (jump height [cm]) + 45.3 × (body mass [kg]) - 2055). Rest intervals will be the amount of time it takes to complete the measurement for each trial.
standing long jump assessment | From enrollment to the end of follow up assessment at 24 hours
  The standing long jump assessment (SLJ) assessment will be performed for five trials with the best performance on the three experimental trials used to determine lower extremity power. The SLJ will be performed like the protocol used by Mann and colleagues with participants performing horizontal jumps as far as they can and measuring the distance from the start point to the back of the subject's backmost heel. The subject must maintain their balance after landing for the trial to be counted. The farthest distance jumped will then be used to calculate power through the regression formula created by Mann and colleagues (Power [W] = 32.49·SLJ [cm] + 39.69·Wt [kg] - 7,608). Rest time between trials will be the amount of time it takes to measure the distance the subject jumped.

CONTACTS AND LOCATIONS:
Locations (1):
- Blatt PE Center, University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sayers SP, Harackiewicz DV, Harman EA, Frykman PN, Rosenstein MT. Cross-validation of three jump power equations. Med Sci Sports Exerc. 1999 Apr;31(4):572-7. doi: 10.1097/00005768-199904000-00013. PMID 10211854
- [Background] Mann JB, Bird M, Signorile JF, Brechue WF, Mayhew JL. Prediction of Anaerobic Power From Standing Long Jump in NCAA Division IA Football Players. J Strength Cond Res. 2021 Jun 1;35(6):1542-1546. doi: 10.1519/JSC.0000000000004043. PMID 33927119
- [Background] Blazevich AJ, Gill ND, Kvorning T, Kay AD, Goh AG, Hilton B, Drinkwater EJ, Behm DG. No Effect of Muscle Stretching within a Full, Dynamic Warm-up on Athletic Performance. Med Sci Sports Exerc. 2018 Jun;50(6):1258-1266. doi: 10.1249/MSS.0000000000001539. PMID 29300214
- [Background] Taber CB, Colter RJ, Davis JJ, Seweje PA, Wilson DP, Foster JZ, Merrigan JJ. The Effects of Body Tempering on Force Production, Flexibility and Muscle Soreness in Collegiate Football Athletes. J Funct Morphol Kinesiol. 2022 Jan 11;7(1):9. doi: 10.3390/jfmk7010009. PMID 35076554
- See also: body tempering devices — https://www.roguefitness.com/rogue-dt-tempering-roller
- See also: body tempering table — https://www.roguefitness.com/dt-tempering-table